CLINICAL TRIAL: NCT07044401
Title: A Phase 1, Randomized, Open-label, Single-Dose, Crossover Study to Investigate the Effect of Injection Site on Relative Bioavailability of KAI-9531 Subcutaneous Injection in Participants With a Range of Body Mass Indices
Brief Title: A Single-dose Study to Investigate the Effect of Injection Site on KAI-9531 Relative Bioavailability in a Range of Body Mass Indices
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kailera (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: K9531-1102
Record Dates: First submitted 2025-06-23; First posted 2025-07-01 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Healthy Volunteers
Keywords: Overweight; Obesity; KAI-9531
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- KAI-9531: Abdomen Injection Site (Experimental): Participants will receive KAI-9531 as a SC injection into the abdomen on Day 1 of either Treatment Period 1, 2 or 3.
  Interventions: Drug: KAI-9531
- KAI-9531: Thigh Injection Site (Experimental): Participants will receive KAI-9531 as a SC injection into the thigh on Day 1 of either Treatment Period 1, 2 or 3.
  Interventions: Drug: KAI-9531
- KAI-9531: Upper Arm Injection Site (Experimental): Participants will receive KAI-9531 as a SC injection into the upper arm on Day 1 of either Treatment Period 1, 2 or 3.
  Interventions: Drug: KAI-9531

INTERVENTIONS:
Drug: KAI-9531 — SC Injection.

SUMMARY:
The main objective of the study is to assess the relative bioavailability of KAI-9531 subcutaneous (SC) injection in the upper arm and thigh compared to the abdomen.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) ≥ 25.0 and ≤ 40.0 kilograms per square meter (kg/m^2), with a body weight ≤ 120 kg.
* Medically healthy.

Exclusion Criteria:

* Known hypersensitivity to the study drug or any of the study drug ingredients.
* History or presence of clinically significant cardiovascular, pulmonary, hepatic, renal, hematological, gastrointestinal, endocrine, immunologic, dermatologic, psychiatric, or neurological disease/disorder.
* Any history of malignant disease in the last 10 years (excludes surgically resected skin squamous cell or basal cell carcinoma).
* Estimated glomerular filtration rate (eGFR) <60 milliliters per minute per 1.73 square meters of body surface area (mL/min/1.73 m^2) using the 2021 Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation.
* Glycosylated hemoglobin (HbA1c) test result ≥6.5%.
* A history of or positive test results at the Screening visit for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV) antibody (HCVab) with HCV ribonucleic acid (RNA) confirmation if positive.
* Positive drugs of abuse or alcohol test results.
* Participation in another clinical study of an investigational drug or investigational device within 30 days or 5 half-lives of the investigational drug (whichever is longer).
* Any other condition or prior therapy that would make the participant unsuitable for this study, including inability to cooperate fully with the requirements of the study protocol or likelihood of noncompliance with any study requirements.

Note: Additional inclusion/exclusion criteria may apply, per protocol.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2025-07-14 (Actual); Primary Completion 2025-11-13 (Actual); Study Completion 2025-11-13 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Concentration (Cmax) of KAI-9531 | Treatment Period 1, 2 and 3: Pre-dose and up to 672 hours post-dose
Area Under the Concentration-time Curve From 0 to Time of Last Quantifiable Concentration (AUC0-t) of KAI-9531 | Treatment Period 1, 2 and 3: Pre-dose and up to 672 hours post-dose
Area Under the Concentration-time Curve From 0 to Infinity (AUC0-inf) of KAI-9531 | Treatment Period 1, 2 and 3: Pre-dose and up to 672 hours post-dose

SECONDARY OUTCOMES:
Number of Participants Who Experience a Treatment-emergent Adverse Event (TEAE) | Day 1 to Day 113
Number of Participants Who Experience a Serious Adverse Event (SAE) | Day 1 to Day 113
Number of Participants Who Experience Antidrug Antibodies to KAI-9531 | Day 1 to Day 113

CONTACTS AND LOCATIONS:
Locations (1):
- Celerion, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: No